CLINICAL TRIAL: NCT06236750
Title: A Post-Marketing Surveillance to Observe the Safety and Efficacy of Dehydrated Human Amnion/Chorion Membrane (DHACM) Wound Graft in the Management of Non-Ischemic Chronic Wounds
Brief Title: Post-Marketing Surveillance of Dehydrated Human Amnion/Chorion Membrane (DHACM) in Non-Ischemic Chronic Wounds
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MiMedx Group, Inc. (Industry)
Collaborators: CMIC Co, Ltd. Japan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EFJP001
Record Dates: First submitted 2024-01-24; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Diabetic Foot Ulcer; Venous Leg Ulcer
MeSH Terms: conditions — Diabetic Foot; Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Non-Ischemic Chronic Wounds (Experimental): Patients with intractable diabetic foot ulcer or venous leg ulcer that have not decreased in surface area by at least 50% after 4 weeks of conventional therapies.
  Interventions: Device: EPIFIX

INTERVENTIONS:
Device: EPIFIX — EPIFIX® is an allograft derived from dehydrated human amnion/chorion membrane. EPIFIX is a medical device in Japan (Generic name: Material using human amniotic membrane for promotion of tissue healing) for use on intractable ulcers that are non-responsive to existing therapies for the purpose of promoting wound healing.
  Other Names: DHACM

SUMMARY:
The purpose of this survey is to observe the efficacy and safety of EPIFIX® dehydrated human amnion/chorion membrane (DHACM) for the treatment of intractable diabetic foot ulcers or venous leg ulcers.

DETAILED DESCRIPTION:
The study will enroll 75 subjects diagnosed with intractable diabetic foot ulcers or venous leg ulcers at 5 plastic surgery sites in Japan. Subjects will be treated with weekly applications of EPIFIX for up to 12 weeks, followed by 6 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

Patients with intractable diabetic foot ulcers or venous leg ulcers that have not decreased in surface area by at least 50% after 4 weeks of conventional therapies, such as radical wound management (removal of necrotic tissue, infection control, wound cleansing, etc.), glycemic control for diabetic foot ulcers, compression therapy for venous stasis ulcers and moist therapy using wound dressing materials.

Exclusion Criteria:

1. Areas of active infection or latent infection.
2. Patients with disorders that would cause an intolerable risk of postoperative complications.
3. Ulcers that cannot be sufficiently debrided.
4. Ulcers that, after debridement, have blood flow disorders where wound bed necrosis progresses at an early stage.
5. Wound surfaces with multiple ulcer surfaces and exposed bone, and no blood flow in the wound bed.
6. Patients with hypersensitivity to the aminoglycoside antibiotics used during manufacturing.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-08-04 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy Endpoint: Healing of Ulcers at 4 Weeks, 8 Weeks, and 12 Weeks | 4 weeks, 8 weeks, and 12 weeks after initial application
  The percentage of patients to achieve wound closure at 4 weeks, 8 weeks, and 12 weeks after initial DHACM application, as a measure of healing rate.
Safety Endpoint: Incidence of Adverse Events | 9 months after initial application
  Incidence rate of adverse events in DHACM-treated patients during 12 weeks of treatment and 6 months of follow-up.

OTHER OUTCOMES:
Efficacy Endpoint: Reduction in Wound Size at 4 Weeks, 8 Weeks, and 12 Weeks | 4 weeks, 8 weeks, and 12 weeks after initial application
  Wound size will be measured at 4 weeks, 8 weeks, and 12 weeks after initial DHACM application, and the percent reduction of wound area will be calculated compared to baseline (week 0), as a measure of rate of wound closure.
Efficacy Endpoint: Time to Complete Wound Healing during 12 Weeks of Application | 12 weeks after initial application
  The amount of time after initial DHACM application to achieve complete epithelialization of the wound.
Efficacy Endpoint: Wound Recurrence for 6 months after Wound Closure | 6 months after wound closure
  The recurrence rate of healed ulcers will be monitored for 6 months after wound closure is achieved.
Safety Endpoint: Incidence of Device Deficiencies | 9 months after initial application
  Incidence rate of device deficiencies, severity, and details in DHACM-treated patients during 12 weeks of treatment and 6 months of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: David Mason, MD, Study Director — MiMedx Group, Inc.
Locations (5):
- Japan (5):
  - Kobe University Hospital, Kobe, Hyōgo
  - Saitame Medical University Hospital, Iruma-gun, Saitama
  - Juntendo University Hospital, Bunkyō-Ku, Tokyo
  - Kyorin University Hospital, Mitaka-shi, Tokyo
  - Tokyo Medical University Hospital, Shinjuku-Ku, Tokyo